CLINICAL TRIAL: NCT03149003
Title: A Randomized, Multicenter, Adaptive Phase 3 Study of DSP-7888 Dosing Emulsion in Combination With Bevacizumab Versus Bevacizumab Alone in Patients With Recurrent or Progressive Glioblastoma Following Initial Therapy (WIZARD 201G)
Brief Title: A Study of DSP-7888 Dosing Emulsion in Combination With Bevacizumab in Patients With Recurrent or Progressive Glioblastoma Following Initial Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI-DSP7888-201G
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2023-01-30 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma
Keywords: Glioblastoma (GBM); Wilms Tumor 1 (WT1); Cancer Vaccines; Neoplasms; Astrocytoma; Glioma; Brain Cancer; Brain Tumor; Bevacizumab
MeSH Terms: conditions — Glioblastoma; Wilms Tumor; Neoplasms; Astrocytoma; Glioma; Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: DSP-7888 Dosing Emulsion plus Bevacizumab (Experimental)
  Interventions: Drug: DSP-7888 Dosing Emulsion; Drug: Bevacizumab
- Arm 2: Bevacizumab (Active Comparator)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: DSP-7888 Dosing Emulsion — DSP-7888 Dosing Emulsion will be administered i.d. every 7 ± 1 day for Doses 1 to 5, every 14 ± 3 days for Doses 6 to 15, and every 28 ± 7 days for Doses 16 and above.
  Other Names: adegramotide and nelatimotide
  Arms: Arm 1: DSP-7888 Dosing Emulsion plus Bevacizumab
Drug: Bevacizumab — Bevacizumab will be administered intravenously every 14 ± 3 days at 10 mg/kg.
  Other Names: Avastin

SUMMARY:
This is an event driven, adaptive design, a randomized, active-controlled, multicenter, open-label, parallel groups, Phase 3 study of DSP-7888 Dosing Emulsion plus Bevacizumab versus Bevacizumab alone in patients with recurrent or progressive glioblastoma multiforme (GBM) following treatment with first line therapy consisting of surgery and radiation with or without chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients or their legal representatives must be able to provide written informed consent.
* Histologically confirmed diagnosis of supratentorial GBM (Grade 4 astrocytoma).
* Radiographic evidence of first recurrence or progression of GBM following primary therapy consisting of surgery (biopsy or resection) and chemoradiation; patients may have undergone a second debulking surgery following initial recurrence or progression. Patients whose tumors are O6 methyl guanyl-methyltransferase (MGMT) methylated-promoter negative need not have received chemotherapy in the past to be eligible.
* Human leukocyte antigen type HLA-A*02:01, HLA-A*02:06, or HLA-A*24:02.
* Age ≥18.
* KPS score of ≥60.
* Serum creatinine value <2X the upper limit of normal (ULN) for the reference laboratory.
* Alanine aminotransferase/aspartate aminotransferase <3X the ULN and total bilirubin <2× the ULN for the reference laboratory.
* Men and women of childbearing potential must agree to use a reliable method of contraception (oral contraceptives, implantable hormonal contraceptives, or double barrier method) or agree to completely refrain from heterosexual intercourse for the duration of the study and for 180 days following the last dose of DSP-7888 Dosing Emulsion.
* Patients must have recovered from the effect of all prior therapy to Grade 2 or less.
* Patients must be at least 28 days from any major surgery, and any surgery incisions or wounds must be completely healed.
* Patients must be at least 12 weeks from the completion of prior radiation therapy (RT) in order to discriminate pseudo progression of disease from progression.
* Patients must be at least 4 weeks from the completion of prior systemic or intracranial chemotherapy.
* Patients must stop Novo-TTF treatment one day prior to study therapy (no washout period is needed). However, any wounds from TTF must be adequately healed per Inclusion Criterion #11.15. For patients who are not receiving therapeutic anticoagulation treatment, an international normalized ratio (INR) and a PTT ≤ 1.5 × the ULN; patients who are receiving anticoagulation treatment should be on a stable dose.
* Patient's left ventricular ejection fraction (LVEF) > 40%. 17. Patient has a resting pulse oximetry of 90% or higher.

Exclusion Criteria:

Patients with any of the following will be excluded from the study:

* Prior therapy with Bev.
* Patients with secondary GBM.
* Any anti-neoplastic therapy, including RT, for first relapse or recurrence.
* Evidence of leptomeningeal spread of tumor or any history, presence, or suspicion of metastatic disease extracranially.
* Evidence of impending herniation on imaging.
* Has known multifocal disease. Multifocal disease is defined as discrete sites of disease without contiguous T2/FLAIR abnormality that require distinct radiotherapy ports. Satellite lesions that are associated with a contiguous area of T2/FLAIR abnormality as the main lesion(s) and that are encompassed within the same radiotherapy port as the main lesion(s) are permitted.
* Patients with infections that have required treatment with systemic antibiotics within 7 days of first dose of protocol therapy.
* The need for systemic glucocorticoids in doses in excess of 4 mg/day of dexamethasone or in comparable doses with other glucocorticoids.
* Treatment with any investigational agents within 5 half-lives of the agent in question or, if the half-life is unknown, within 28 days of enrollment.
* Pregnant or lactating females.
* Prior history of malignancy within 3 years of enrollment other than basal or squamous cell carcinoma of the skin, cervical intra-epithelial neoplasia, in situ carcinoma of the breast, or prostate cancer treated with surgery or RT with a prostate specific antigen of <0.01 ng/mL.
* Patients with active autoimmune diseases within 2 years of enrollment into the study including, but not limited to, rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, Sjogren's syndrome, Wegener's granulomatosis, ulcerative colitis, Crohn's disease, myasthenia gravis, Graves' disease, or uveitis except for psoriasis not requiring systemic therapy, vitiligo or alopecia areata, or hypothyroidism; if an autoimmune condition has been clinically silent for 12 months or greater, the patient may be eligible for enrollment.
* Patients on immunosuppressive therapies; the use of topical, inhalational, ophthalmologic or intra articular glucocorticoids, or the use of physiologic replacement doses of glucocorticoids are permitted.
* Patients with primary immunodeficiency diseases.
* Patients with significant bleeding in the preceding 6 months or with known coagulopathies.
* History of abdominal fistula, intestinal perforation, or intra-abdominal abscess in the preceding 12 months.
* Positive serology for human immunodeficiency virus (HIV) infection, active hepatitis B*, or untreated hepatitis C; patients who have completed a course of anti-viral treatment for hepatitis C are eligible.

  o *In cases of negative results for HepB surface antigen with positive HepB core antibody, HBV DNA testing is required.
* Patient has a medical history of frequent ventricular ectopy, e.g., non-sustained ventricular tachycardia (VT).
* Significant cardiovascular disease, including New York Hospital Association Class III or IV congestive heart failure, myocardial infarction within 6 months of enrollment, unstable angina, poorly controlled cardiac arrhythmias, or stroke within the preceding 6 months.
* Any other uncontrolled inter current medical condition, including systemic fungal, bacterial, or viral infection; uncontrolled hypertension; diabetes mellitus; or chronic obstructive pulmonary disease requiring 2 or more hospitalizations in the preceding 12 months.
* Any psychiatric condition, substance abuse disorder, or social situation that would interfere with a patient's cooperation with the requirements of the study.
* Known sensitivity to Bev or any of the components of DSP-7888 Dosing Emulsion.
* Patient has a QTcF (QT corrected based on Fridericia's equation) interval > 480 msec (CTCAE = Grade 2) or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) at screening. (Patients with bundle branch block and a prolonged QTc interval should be reviewed by the Medical Monitor for potential inclusion.)
* Patient has dyspnea at rest (CTCAE ≥ Grade 3) or has required supplemental oxygen within 2 weeks of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (37):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Center for Neurosciences, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - UCSD- Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Neuro-Oncology/ US Irvine Medical Center, Orange, California
  - Sansum Clinic, Santa Barbara, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Piedmont brain tumor center, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kentucky / Department of Internal Medicine / Markey Cancer Center, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York
  - Weill Cornell Medicine, New York, New York
  - Columbia University Medical Center/ Neurological Institute of NY, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee Academic Medical Center Cancer Institute, Knoxville, Tennessee
  - Texas Oncology Austin Midtown, Austin, Texas
  - Baylor Scott and White, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - Mischer Neuroscience Associates/Memorial Hermann Hospital, Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin Hospital, Madison, Wisconsin
- Canada (3):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - University of Sherbrooke, Sherbrooke, Quebec
- Japan (12):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Niigata University Medical and Dental Hospital, Chuo Ku, Niigata
  - Osaka International Cancer Institute, Chuo Ku, Osaka
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Kumamoto University Hospital, Kumamoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku
  - Yamagata University Hospital, Yamagata
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab: Drug: DSP-7888 Dosing Emulsion DSP-7888 Dosing Emulsion will be administered i.d. every 7 ± 1 day for Doses 1 to 5, every 14 ± 3 days for Doses 6 to 15, and every 28 ± 7 days for Doses 16 and above.
  Other Name: adegramotide and nelatimotide
  Drug: Bevacizumab Bevacizumab will be administered intravenously every 14 ± 3 days at 10 mg/kg. Other Name: Avastin
- Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab: DSP-7888 Dosing Emulsion: DSP-7888 Dosing Emulsion will be administered i.d. every 7 ± 1 day for Doses 1 to 5, every 14 ± 3 days for Doses 6 to 15, and every 28 ± 7 days for Doses 16 and above.
  Bevacizumab: Bevacizumab will be administered intravenously every 14 ± 3 days at 10 mg/kg.
- Part 2 - Arm 2: Bevacizumab: Bevacizumab: Bevacizumab will be administered intravenously every 14 ± 3 days at 10 mg/kg.
Period: Overall Study
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab
Started | 4 | 109 | 108
Completed | 4 | 108 | 90
Not Completed | 0 | 1 | 18
Not completed — Randomized but not treated | 0 | 1 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab | Total
Number analyzed (Participants) | 4 | 109 | 108 | 221
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 76 | 74 | 153
  >=65 years | 1 | 33 | 34 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 37 | 45 | 85
  Male | 1 | 72 | 63 | 136
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native Aboriginal (including First Nations, Metis, Inuit) | 0 | 0 | 0 | 0
  Caucasian | 3 | 63 | 67 | 133
  Asian | 0 | 38 | 36 | 74
  Black (including African, Caribbean descent) | 0 | 1 | 1 | 2
  Native Americans or Alaskan Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 1 | 7 | 4 | 12
HLA Class I Type [Count of Participants; unit: Participants]
  HLA-A*02 Positive Only | 4 | 67 | 61 | 132
  HLA-A*24 Positive Only | 0 | 29 | 39 | 68
  Both Positive | 0 | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity
Description: The number of participants with dose-limiting toxicity (DLT) who were enrolled into Part 1 - the safety set.
Time Frame: Dose-limiting toxicity will be evaluated and applied from Day 1 through Day 29
Population: Analysis limited to patients enrolled into Part 1 - the safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab
Number analyzed (Participants) | 4 | 0 | 0
Participants | 0 |  |

2. Primary Outcome: Overall Survival (OS) of Patients With Recurrent or Progressive Glioblastoma Multiforme (GBM) Treated With DSP-7888 Dosing Emulsion Plus Bevacizumab (BEV) Versus BEV Alone
Description: The effect of DSP-7888 Dosing Emulsion plus BEV versus BEV alone on the OS of patients with recurrent or progressive GBM following treatment with first line therapy consisting of surgery and radiation with or without chemotherapy.
Time Frame: 4 weeks after the patient has been off study treatment, every 3 months thereafter until death, the study closes, up to 24 months.
Population: Analysis limited to patients randomized into Part 2 - the intent-to-treat set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab
Number analyzed (Participants) | 0 | 109 | 108
months |  | 10.2 [8.2 to 11.4] | 9.4 [7.4 to 10.3]

3. Secondary Outcome: Overall Survival (OS) of Patients With Recurrent or Progressive Glioblastoma Multiforme (GBM) Treated With DSP-7888 Dosing Emulsion Plus Bevacizumab (BEV) Versus BEV Alone at 12 Months
Description: as for outcome 2
Time Frame: 12 months
Population: Analysis limited to patients randomized into Part 2 - the intent-to-treat set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab
Number analyzed (Participants) | 0 | 109 | 108
percentage of participants |  | 37.9 [28.7 to 47.0] | 31.6 [22.9 to 40.7]

4. Secondary Outcome: Progression Free Survival (PFS) of Patients With Recurrent or Progressive GBM
Description: The effect of DSP-7888 dosing emulsion plus Bevacizumab (BEV) versus BEV alone on the Progression Free Survival (PFS) of patients with recurrent or progressive GBM following treatment with first line therapy consisting of surgery and radiation with or without chemotherapy. PFS is defined as the interval between randomization and progression or death from any cause any cause as determined by the central radiology body.
Time Frame: The time from the date of first treatment to the date of first documentation of disease progression or death due to any cause, up to 24 months
Population: Analysis limited to patients randomized into Part 2 - the intent-to-treat set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab
Number analyzed (Participants) | 0 | 109 | 108
months |  | 5.3 [3.9 to 5.6] | 3.8 [3.7 to 5.6]

5. Secondary Outcome: Progression Free Survival (PFS) Rate in Patients With Recurrent or Progressive GBM at 6 Months
Description: The effect of DSP-7888 dosing emulsion plus Bevacizumab (BEV) versus BEV alone on the Progression Free Survival (PFS) rate in patients with recurrent or progressive GBM following treatment with first line therapy consisting of surgery and radiation with or without chemotherapy. PFS is defined as the interval between randomization date and progression or death from any cause as determined by the central radiology body. The percentage of patients who achieved PFS at 6 months are summarized.
Time Frame: The time from the date of first treatment to the date of first documentation of disease progression or death due to any cause at 6 months
Population: Analysis limited to patients randomized into Part 2 - the intent-to-treat set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab
Number analyzed (Participants) | 0 | 109 | 108
percentage of participants |  | 36.3 [26.7 to 46.0] | 35.4 [24.0 to 47.0]

6. Secondary Outcome: The Effect of DSP-7888 Dosing Emulsion Plus Bevacizumab (BEV) Versus BEV Alone on the Response Rate of Patients With Recurrent or Progressive GBM
Description: Assessment of the objective response rate (ORR) of DSP-7888 dosing emulsion plus BEV versus BEV alone in patients with recurrent or progressive GBM. The response rate is defined as the percentage of patients exhibiting a response (complete response [CR] plus partial response [PR]) based on the Modified Response Assessment in Neuro-Oncology (RANO) criteria as determined by the central radiology body.
Time Frame: From the date of first treatment, every 8 weeks, until the date of first documented objective disease progression, up to 24 months
Population: Analysis limited to patients randomized into Part 2 - the intent-to-treat set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab
Number analyzed (Participants) | 0 | 109 | 108
percentage of participants |  | 21.1 [13.9 to 30.0] | 13.0 [7.3 to 20.8]

7. Secondary Outcome: Duration of Response in Patients With Recurrent or Progressive GBM Treated With DSP-7888 Dosing Emulsion Plus Bevacizumab (BEV) Versus BEV Alone
Description: The effect of DSP-7888 dosing emulsion plus BEV versus BEV alone on the duration of response of patients with recurrent or progressive GBM. The duration of response is defined as the interval between first documented oncological response and progression of disease or death from any cause.
Time Frame: From the date of first treatment up to 24 months
Population: Analysis limited to patients randomized into Part 2 - the intent-to-treat set. NE signifies "Not Estimable" in the results.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab
Number analyzed (Participants) | 0 | 109 | 108
months |  | 4.81 (7.119) | 3.69 (4.017)

8. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Assessment of safety of DSP7888 dosing emulsion plus Bevacizumab (BEV) versus BEV alone in patients with recurrent or progressive GBM
Time Frame: The time from the date of first treatment, while the patient is on treatment, and for 30 days after stopping therapy, an average of 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab
Number analyzed (Participants) | 4 | 109 | 108
Participants | 4 | 106 | 79

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed from the date of first treatment through 30 days of the last administration of study drug, an average of 4 months. All-Cause Mortality was assessed from the date of first treatment until death, up to 24 months.
Description: In part 2 of the trial, 109 patients were randomized to arm 1, however 1 patient did not receive study drug and did not complete the trial. Therefore, the 108 patients in arm 1 who were randomized and received study drug were at risk for AEs or SAEs. In part 2 - arm 2, 108 patients were randomized, however 18 patients did not receive study drug and did not complete the trial. Therefore, the 90 patients in arm 2 who were randomized and received study drug were at risk for AEs or SAEs.
Arm/Group | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab | Part 2 - Arm 2: Bevacizumab
All-Cause Mortality (participants affected / at risk) | 4/4 | 96/109 | 89/108
Serious Adverse Events (participants affected / at risk) | 1/4 | 10/108 | 6/90
Other Adverse Events (participants affected / at risk) | 4/4 | 106/108 | 79/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab (N=4) | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab (N=108) | Part 2 - Arm 2: Bevacizumab (N=90)
Seizure (Nervous system disorders) | 1 | 6 | 5
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 2 | 1
Hydrocephalus (Nervous system disorders) | 0 | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 4 | 0
Gait disturbance (General disorders) | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 1 | 0
Putamen haemorrhage (Nervous system disorders) | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0
Wound infection pseudomonas (Infections and infestations) | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab (N=4) | Part 2 - Arm 1: DSP-7888 Dosing Emulsion Plus Bevacizumab (N=108) | Part 2 - Arm 2: Bevacizumab (N=90)
Vomiting (Gastrointestinal disorders) | 2 | 15 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 12 | 11
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 13 | 15
Injection site reaction (General disorders) | 3 | 88 | 0
Fatigue (General disorders) | 2 | 32 | 17
Pyrexia (General disorders) | 2 | 14 | 7
Injection site erythema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 8 | 5
Headache (Nervous system disorders) | 2 | 39 | 23
Seizure (Nervous system disorders) | 2 | 22 | 10
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 6 | 7
Hemiparesis (Nervous system disorders) | 1 | 10 | 8
Decreased appetite (Metabolism and nutrition disorders) | 2 | 14 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Anxiety (Psychiatric disorders) | 1 | 5 | 7
Confusional state (Psychiatric disorders) | 1 | 15 | 6
Insomnia (Psychiatric disorders) | 1 | 10 | 9
Mental status changes (Psychiatric disorders) | 1 | 1 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 15 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 5
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Hyperacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 40 | 24
Gait disturbance (General disorders) | 0 | 10 | 8
Asthenia (General disorders) | 0 | 6 | 5
Aphasia (Nervous system disorders) | 0 | 16 | 11
Memory impairment (Nervous system disorders) | 0 | 10 | 4
Constipation (Gastrointestinal disorders) | 0 | 22 | 11
Abdominal pain (Gastrointestinal disorders) | 0 | 7 | 2
Urinary tract infection (Infections and infestations) | 0 | 15 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 12 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 10 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 9 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 8 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 7 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 6 | 7
Depression (Psychiatric disorders) | 0 | 8 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 9 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 7 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 5 | 6
Proteinuria (Renal and urinary disorders) | 0 | 19 | 9
Urinary incontinence (Renal and urinary disorders) | 0 | 7 | 1
Weight decreased (Investigations) | 0 | 10 | 3
Lymphocyte count decreased (Investigations) | 0 | 8 | 2
Alanine aminotransferase increased (Investigations) | 0 | 7 | 9
Aspartate aminotransferase increased (Investigations) | 0 | 6 | 6
Weight increased (Investigations) | 0 | 5 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 20 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution shall submit to Sponsor for its review a copy of any proposed publication resulting from the study at least thirty days prior to the date of submission for publication. Sponsor shall complete its review within thirty days of its receipt of the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT03149003/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03149003/SAP_001.pdf